CLINICAL TRIAL: NCT05980143
Title: Can Metacognitive Therapy be Used to Treat Common Mental Health Problems in Autistic Children and Adolescents: A Systematic Case Series
Brief Title: Metacognitive Therapy for Common Mental Health Problems in Autistic CYP: A Case Series
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government); Pennine Care NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Adrian Wells, Professor, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 320925
Record Dates: First submitted 2023-05-09; First posted 2023-08-07 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Depression
Keywords: Anxiety symptoms; Depression symptoms; Metacognitive therapy; Children and young people; Autism
MeSH Terms: conditions — Anxiety Disorders; Depression; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metacognitive Therapy (Experimental): MCT will be delivered in accordance with the MCT-PATHWAY treatment manual.
  Interventions: Other: Metacognitive Therapy

INTERVENTIONS:
Other: Metacognitive Therapy — The transdiagnostic Metacognitive model suggests that psychological difficulties arise from the activation of a thinking style called the CAS (Cognitive Attentional Syndrome). Metacognitive Therapy (MCT) aims to bring the CAS under control. The therapist helps the patient to learn new ways of relating to stressful thoughts.

SUMMARY:
Anxiety and Depression are common in young people (CYP) and especially in CYP with a diagnosis of Autism. Autistic people often say therapy has not been adapted to meet their needs. A recent treatment called metacognitive therapy (MCT) is proving to be helpful, but the investigators do not know how autistic CYP will find MCT, or what changes to the delivery of therapy may be needed to meet their needs. This study hopes to explore whether MCT can help treat anxiety and/or depression in autistic young people.

This study aims to offer five autistic CYP MCT. To take part, they must be between 11-16 years old and have depression and/or anxiety symptoms. The study will involve completing questionnaires at the start, during therapy, at the end and after 6 months. Therapy will be scheduled for at least eight sessions. Therapy involves working on what we think about our worry, rather than on specific worries. What we think about our worry can be positive or negative. For example, 'worrying helps me cope' and 'worrying could make me go mad'. This can affect where our attention goes and how we think. At the end of therapy, participants will be asked to take part in an interview about how they found the therapy.

The questionnaires will help test how useful the measures are, suggest how helpful the therapy might be and whether benefits continue after the therapy has ended. Information will also be gathered through a post treatment interview about how the young people found the therapy. This will help understand whether any changes to the therapy are needed to meet the needs of autistic people. This information is necessary for planning a large-scale trial for autistic CYP. Such studies may improve treatment options and service provision for mental health problems in this population.

Primary Question:

• Is MCT a feasible and acceptable treatment for treating anxiety and depression in autistic CYP?

Secondary Questions:

* Is MCT associated with clinically significant change in outcome measures following the introduction of treatment for autistic CYP?
* Are improvements associated with MCT maintained at 6 month follow up?
* Are improvements associated with MCT replicable across autistic CYP?
* Do the investigators need to modify how MCT is delivered to autistic CYP?

DETAILED DESCRIPTION:
This study is a systematic replication case series utilising an AB design with follow up to deliver MCT to autistic CYP who experience symptoms of anxiety and/or depression. Allocation to baseline lengths will not be randomised, natural baselines will be utilised whereby participants complete the primary outcome measure weekly until they demonstrate stability. Stability will be defined as an absence of decreasing trend of at least three consecutive data points prior to the introduction of treatment.

Recruitment:

Participants will be identified by CAMHS clinicians during routine clinical practice. Potential participants will be provided with information about the study, including the participant information sheet. Those who are identified as eligible and are interested in taking part or finding out more about the study will consent to their details being shared with the researcher. The details will be securely sent to the researcher using the eligibility form. The researcher will then contact potential participants to confirm whether the like to participate and answer any questions they have about the study.

Screening:

Those who wish to participate will then be invited to attend a screening appointment with the researcher. Written consent will be obtained from participants (and parents/guardians where appropriate). Once consent has been obtained, demographic information, baseline measures will be administered.

Baseline:

During the baseline phase, participants will be asked to complete the Personal Rating Scale and the YoCas-1 once a week for a minimum of 3 weeks, until stability is achieved. Only the Personal Rating Scale will be used to measure stability. Stability is defined as the absence of a decreasing trend on three consecutive data points prior to the introduction of treatment. All other outcome measures will be completed at the end of the baseline phase prior to starting treatment.

Intervention:

Participants will be offered a minimum of eight weekly sessions of MCT at their local CAMHS. Each session will last approximately an hour. This will be applied flexibly, and sessions can be extended in response to client progress. This will provide information about whether the investigators need to modify the delivery of MCT to autistic CYP. Participants will be asked to complete sessional measures.

Post Intervention interview:

Participants will be asked to take part in the post intervention interview to gather information about how they found the intervention. This will consider factors such as components of the intervention that were well received, and those which were less well received.

Follow up:

Participants will be asked to complete follow up measures 6 months after the final treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Age between 11-16 years
* Consent given
* Formal diagnosis of Autism Spectrum Disorder
* Fluent in English
* Seeking treatment for emotional disorder symptoms (i.e., generalised anxiety disorder, panic disorder, agoraphobia, post-traumatic stress disorder, obsessive compulsive disorder, social anxiety; and/or depression)
* Medication for mental health problems permitted but participants must be stabilised for 6 weeks

Exclusion Criteria:

* Presence of significant risk or safeguarding concerns
* Head injury/organic impairment
* Attention Deficit Hyperactivity Disorder (formal diagnosis or under assessment)
* Eating Disorder

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change in The Revised Children's Anxiety and Depression Scale (RCADS-25) Score | Baseline period: baseline time one to end of baseline, 4-6 weeks post baseline; end of treatment:12-16 weeks post-baseline one; and 6 month follow up.
  A 25-item screening measure designed to assess anxiety and depressive disorders in CYP aged 8-18.
  Anxiety (15 items; maximum score 45) and depression (10 items; maximum score = 30).
  In response to each item, participants must select the appropriate response from 'Always' (score = 3), 'Often' (score = 2), 'Sometimes' (score = 1), 'Never' (score = 0).
  Total minimum score = 0. Total maximum score = 75. Higher scores indicate worse outcomes.
Measure of Credibility and Expectancy | Intervention session 1 (3-6 weeks after 1st baseline measure, dependant on length of baseline)
  A 3 item measure developed by the researchers measuring expectancy and credibility on a 10 point scale
Measure of Adherence and User Friendliness | Final intervention session (12-16 weeks post baseline dependent on whether sessions are extended in response to participant needs)
  A 5 item measure developed by the researchers to measure adherence and user friendliness on a 10 point scale
Post Intervention Interview | 12-16 weeks post baseline (dependent on whether sessions are extended in response to participant needs)
  A semi structured interview focusing on perceived benefits and challenges of the therapy, as well as specific aspects of the therapy such as the outcome measures or intervention techniques.
Change in Personal Rating Scale Score | Weekly during baseline and intervention (across 12-16 weeks dependant on length of baseline and intervention) and at 6 months follow up)
  A personal rating scale developed by the researchers, to be administered weekly measuring how distressing the problem has been and how much the problem has interfered with day to day life

SECONDARY OUTCOMES:
Change in The Youth Cognitive Attentional Syndrome-1 (YoCAS-1) Score | Weekly during baseline and intervention (across 12-16 weeks dependant on length of baseline and intervention) and at 6 months follow up)
  A 7 item self-report measure to assess metacognitive skills and knowledge in youth, including worry/rumination, threat monitoring, coping behaviours and metacognitive beliefs.
Change in Metacognitions Questionnaire - Adolescent version (MCQ-A) Score | Baseline period: baseline time one and at end of baseline, 4-6 weeks post baseline; end of treatment: at 12-16 weeks post-baseline one; and 6 month follow up.
  A 30-item scale designed to measure metacognitive beliefs in adolescents.
Change in Child Health Utility -9D (CHU-9D) Score | Baseline period: baseline time one and at end of baseline, 4-6 weeks post baseline; end of treatment: at 12-16 weeks post-baseline one; and 6 month follow up.
  A 9 item self-report questionnaire to assess health related quality of life in 7-17-year-olds.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Manchester University NHS Foundation Trust, Manchester
  - Pennine Care NHS Foundation Trust, Manchester

REFERENCES:
- [Background] Ebesutani C, Reise SP, Chorpita BF, Ale C, Regan J, Young J, Higa-McMillan C, Weisz JR. The Revised Child Anxiety and Depression Scale-Short Version: scale reduction via exploratory bifactor modeling of the broad anxiety factor. Psychol Assess. 2012 Dec;24(4):833-45. doi: 10.1037/a0027283. Epub 2012 Feb 13. PMID 22329531
- [Background] Cartwright-Hatton S, Mather A, Illingworth V, Brocki J, Harrington R, Wells A. Development and preliminary validation of the Meta-cognitions Questionnaire-Adolescent Version. J Anxiety Disord. 2004;18(3):411-22. doi: 10.1016/S0887-6185(02)00294-3. PMID 15125986
- [Background] Stevens K. Valuation of the Child Health Utility 9D Index. Pharmacoeconomics. 2012 Aug 1;30(8):729-47. doi: 10.2165/11599120-000000000-00000. PMID 22788262
- [Background] Wells, A. (2009). Metacognitive Therapy for Anxiety and Depression. New York: Guilford Press
- [Background] Wells A, Matthews G. Modelling cognition in emotional disorder: the S-REF model. Behav Res Ther. 1996 Nov-Dec;34(11-12):881-8. doi: 10.1016/s0005-7967(96)00050-2. PMID 8990539
- [Background] Wells A. Breaking the Cybernetic Code: Understanding and Treating the Human Metacognitive Control System to Enhance Mental Health. Front Psychol. 2019 Dec 12;10:2621. doi: 10.3389/fpsyg.2019.02621. eCollection 2019. PMID 31920769
- [Background] Simonoff E, Pickles A, Charman T, Chandler S, Loucas T, Baird G. Psychiatric disorders in children with autism spectrum disorders: prevalence, comorbidity, and associated factors in a population-derived sample. J Am Acad Child Adolesc Psychiatry. 2008 Aug;47(8):921-9. doi: 10.1097/CHI.0b013e318179964f. PMID 18645422
- [Background] Normann N, Morina N. The Efficacy of Metacognitive Therapy: A Systematic Review and Meta-Analysis. Front Psychol. 2018 Nov 14;9:2211. doi: 10.3389/fpsyg.2018.02211. eCollection 2018. PMID 30487770
- [Background] Cooper K, Loades ME, Russell AJ. Adapting Psychological Therapies for Autism - Therapist Experience, Skills and Confidence. Res Autism Spectr Disord. 2018 Jan 1;45:43-50. doi: 10.1016/j.rasd.2017.11.002. PMID 30245739
- [Background] Barlow, D. H., Nock, M., & Hersen, M. (2008). Single case research designs: Strategies for studying behaviour change.